CLINICAL TRIAL: NCT01730300
Title: Genitourinary Symptoms in Women Using Levonorgestrel Releasing Intrauterine Systems
Brief Title: Genitourinary Symptoms With Levonorgestrel Releasing Intrauterine Systems
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, murat ekin, Training Officer of Obstetrics and Gynecology Department M.D., Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: LN-IUSBDSK
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main purpose of the study was to evaluate the efficacy of Levonorgestrel Releasing Intrauterine devices (LNR-IUD) on genitourinary symptoms in patients with abnormal uterine bleeding. The patients were asked urogenital distress inventory (UDI) (which includes; irritative symptoms, stress symptoms, obstructive discomfort) and incontinence impact questionnaire (IIQ) (which includes; physical activity, travel, social/relationships, emotional health)questionnaires in the day of application LNR-IUD and six months later this procedure. Statistical analyse will be performed to evaluate the changes in this time period.

ELIGIBILITY:
Inclusion Criteria:

* women using levonorgestrel releasing intrauterine device for the treatment of menorrhagia or adenomyosis

Exclusion Criteria:

* none

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 15-55 aged women using levonorgestrel releasing intrauterine device for the treatment of menorrhagia or adenomyosis
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Urinary frequency | 6 months
  We think that the urinary frequency will be lesser after 6 months of the therapy.

SECONDARY OUTCOMES:
social activity | 6 months
  We think that social activity will be better after reducing urinary symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Murat Ekin, M.D., Study Chair — Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Department of Obstetrics and Gynecology; Cihan Kaya, M.D., Principal Investigator — Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Department of Obstetrics and Gynecology; Mehmet E Ayag, M.D., Principal Investigator — Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Department of Obstetrics and Gynecology
Locations (1):
- Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Department of Obstetrics and Gynecology, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Ekin M, Cengiz H, Ayag ME, Kaya C, Yasar L, Savan K. Effects of the levonorgestrel-releasing intrauterine system on urinary symptoms in patients with adenomyosis. Eur J Obstet Gynecol Reprod Biol. 2013 Oct;170(2):517-20. doi: 10.1016/j.ejogrb.2013.07.019. Epub 2013 Aug 3. PMID 23916583